CLINICAL TRIAL: NCT04544358
Title: iBAILA - Investigating Brains & Activity to Improve Latino Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Xavier Marquez, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0497
Record Dates: First submitted 2020-08-31; First posted 2020-09-10 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Behavior; Cognitive Impairment
MeSH Terms: conditions — Sedentary Behavior; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Random assignment to intervention (BAILAMOS program) or control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAILAMOS© (Experimental): BAILAMOS© includes a 4-month, twice-weekly dance program. The PI and a professional dance instructor co-developed an extensive BAILAMOS© Dance Manual and class-by-class schedule.
  Interventions: Behavioral: BAILAMOS©
- Control (No Intervention): Randomized to wait list, received BAILAMOS© program after data collection.

INTERVENTIONS:
Behavioral: BAILAMOS© — BAILAMOS© includes a 4-month, twice-weekly dance program. The PI and a professional dance instructor co-developed an extensive BAILAMOS© Dance Manual and class-by-class schedule.
  Arms: BAILAMOS©

SUMMARY:
Examine the impact of the BAILAMOS (TM) dance program on lifestyle physical activity

DETAILED DESCRIPTION:
Examine the impact of the BAILAMOS (TM) dance program on lifestyle physical activity (PA). Hypothesis 1: Intervention group will demonstrate greater improvement in Lifestyle PA than controls. 2) Test the impact of BAILAMOS (TM) on cognitive function and quality of life. Hypothesis 2: Intervention group will demonstrate greater improvement in cognitive function and quality of life than controls. 3) Test the impact of BAILAMOS (TM) on brain network functional connectivity. Hypothesis 3: Intervention group will demonstrate enhanced Default Mode Network (DMN), Executive Network (EN), and sensorimotor network connectivity vis a vis controls.

ELIGIBILITY:
Inclusion Criteria:

* age > 60 years;
* Latino/Hispanic;
* ability to speak Spanish;
* participation in <150 minutes/week of aerobic exercise;
* adequate cognitive status as assessed by the Mini Mental State Examination (>14/21);
* danced < 2 times/month over the past 12 months;
* willingness to be randomly assigned to treatment or control group;
* no plans to leave the U.S. > two weeks during the study.

Exclusion Criteria:

* uncontrolled cardiovascular disease or diabetes mellitus;
* pacemaker or metallic implants (infusion pumps, metal prostheses, metallic-backed transdermal patches or metallic shrapnel); - claustrophobia that precludes MRI;
* stroke within the past year;
* healing or unhealed fracture(s);
* hip or knee replacement within the past 6 months;
* heart failure;
* recurrent falls within the past year;
* regular use of a walker or wheelchair;
* weigh more than 300 pounds, as unable to fit into MRI. The EASY (Resnick et al., 2008) will be used to learn if physician consent is needed for program enrollment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David X Marquez, PhD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BAILAMOS© | Control
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAILAMOS© | Control | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (6.02) | 66.8 (7.18) | 67.18 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire for Older Adults
Description: Report minutes of moderate to vigorous level physical activity per week. Weekly frequency and duration of physical activity is used to calculate minutes of moderate to vigorous level physical activity (MVPA) per week.
Time Frame: Baseline and 4 months (follow up) .The 4-month post-intervention follow-up assesses average physical activity over the past 4 weeks.
Population: Only participants that provided data are analyzed.
Measure: Mean (Standard Deviation); unit: Minutes per week
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Minutes per week
  Baseline Total Leisure PA | 402.0 (364.8) | 315.0 (287.2)
  Follow-up Total Leisure PA | 492.0 (241.8) | 326.3 (218.5)

2. Primary Outcome: Activity Counts Per Minute (CPM).
Description: Measured through a wrist-worn accelerometer (ActiGraph Model GT3X) worn for 7 days.
Time Frame: Baseline and 4 months (follow up)
Population: Complete data (pre and post) for treatment group and control group were analyzed and are presented here.
Measure: Mean (Standard Deviation); unit: Counts per Minute (CPM) per day
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 5
Counts per Minute (CPM) per day
  CPM per day Baseline | 13,564.14 (3274.16) | 13,403.02 (2,967.07)
  CPM per day Follow-up | 13,765.39 (3078.331) | 14,431.7 (3,916.80)

3. Secondary Outcome: Trail Making Test (TMT) Part A
Description: Measure of executive function. In part A, the subject connects a series of encircled numbers in numerical order. In part B, the subject connects encircled numbers and letters in numerical and alphabetical order, alternating between the numbers and letters. TMT score is the time in seconds it takes the subject to complete the test. A lower score/time is better. TMT A scores range from 0-180 seconds and TMT B scores range from 0-300 seconds. Raw scores were converted to z-scores utilizing baseline means and standard deviations. Z-scores were then combined into composite scores of executive function.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
Seconds | -1.67 [-15.68 to 12.35] | -18.20 [-44.80 to 8.41]

4. Secondary Outcome: Stroop C (Color)
Description: Measure of executive function. The Stroop test assesses the ability to inhibit cognitive interference. Color-words are printed in inconsistent color ink. Subjects are asked to name the color of the ink and not read the word. Score range is the number of words named correctly minus errors in 30 seconds and ranges from 0-77. Higher scores reflect better performance and less interference on reading ability. Raw scores were converted to z-scores utilizing baseline means and standard deviations. Z-scores were then combined into composite scores of executive function.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
words | -7.00 [-13.52 to -0.47] | -0.20 [-12.09 to 11.69]

5. Secondary Outcome: Stroop C-W (Color-word Test) of the Stroop Neuropsychological Screening Test
Description: as for outcome 4
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
words | -2.42 [-6.56 to 1.72] | 0.80 [-6.46 to 8.06]

6. Secondary Outcome: Verbal Fluency Test - Animals
Description: This is a widely used measure of verbal fluency (or semantic memory) in which the participant is asked to generate exemplars of each of two categories (animals, fruits and vegetables) within a 60-second time limit. The primary measure of performance is the number of unique exemplars generated within the time limit. The score is the total number of animals (Animal Total) and vegetables (Vegetable Total) named within the time limit. A higher score means a better outcome. Scores range from 0 with no upper limit.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
words | -0.67 [-3.11 to 1.78] | 1.00 [0.12 to 1.88]

7. Secondary Outcome: Symbol Digit Modalities Test
Description: Measure of the speed of perceptual processing in which the participant is asked to identify and name the numbers which belong with consecutively presented symbols for 90 seconds. The score is the number of digits correctly identified within the 90-second time limit - a higher score means a better outcome. Scores range from 0 to 110.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: symbols
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
symbols | 2.17 [0.79 to 3.54] | 4.20 [2.36 to 6.04]

8. Secondary Outcome: Digit Span Test - Forward
Description: This is a widely used measure of working memory (or attention) in which the participant is read number sequences of increasing length and then asked to repeat each sequence forward (Digits Forward) or backward (Digits Backward). The primary measure of performance is the number of digit sequences correctly recalled in each subpart (Digits Forward, Digits Backward). Each sequence for Digits Forward and Digits Backward is scored as error (0) or correct (1) - a higher score means a better outcome.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
score on a scale | 0.25 [-0.93 to 1.43] | -0.20 [-1.24 to 0.84]

9. Secondary Outcome: Digit Ordering Test
Description: This is a measure of working memory in which the participant is read number sequences of increasing length and is then asked to reorder the digits and say them in ascending order. Score range is 0 - 12 with a higher score meaning a better outcome.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
score on a scale | 0.17 [-0.73 to 10.6] | 1.40 [-0.48 to 3.28]

10. Secondary Outcome: Logical Memory I (Immediate) Test
Description: Measure This is a measure of memory (declarative/episodic) in which a brief story is read to P who is then asked to retell it from memory immediately (I) and after a delay (II). The primary measure of performance is the number of story units recalled. Score is the sum of story units (25) correctly recalled. Scores range from 0 - 25 with a higher score meaning a better outcome.
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
score on a scale | -0.08 [-1.42 to 1.26] | 1.00 [-1.92 to 3.92]

11. Secondary Outcome: Logical Memory II (Delayed) Test
Description: as for outcome 10
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
score on a scale | -0.83 [-2.10 to 0.43] | 1.40 [0.72 to 2.08]

12. Secondary Outcome: Cerebral White Matter Volume - Global
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 417,408.33 (64,053.55) | 405,458.70 (41,940.88)

13. Secondary Outcome: Cerebral White Matter Volume - Frontal
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 130,416.27 (21,216.58) | 128,372.50 (11,343.96)

14. Secondary Outcome: Cerebral White Matter Volume - Temporal
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 38,062.08 (6,461.32) | 37,748.52 (4,514.79)

15. Secondary Outcome: Cerebral White Matter Volume - Parietal
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 67,813.37 (10,123.13) | 68,110.53 (7,466.84)

16. Secondary Outcome: Cerebral White Matter Volume - Occipital
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 42,533.23 (5,397.18) | 40,715.26 (5,742.96)

17. Secondary Outcome: Cerebral White Matter Volume - Anterior Cingulate
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 9,596.52 (1,595.92) | 9,099.53 (618.19)

18. Secondary Outcome: Cerebral White Matter Volume - Posterior Cingulate
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline and 4 months (follow up)
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 8,326.62 (1,210.24) | 7,850.10 (874.68)

19. Secondary Outcome: Cerebral White Matter Volume - Isthmus of the Cingulate
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 6,578.39 (1,091.53) | 6,625.83 (685.92)

20. Secondary Outcome: Cerebral White Matter Hyper-intensities
Description: Assessed through magnetic resonance imaging scans
Time Frame: Baseline
Population: A subsample of 14 participants participated in MRI scans. We analyzed and published baseline data for this outcome.
Measure: Mean (Standard Deviation); unit: Cubic millimeters
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 4
Cubic millimeters | 1728.66 (1194.1) | 2567.49 (782.40)

21. Secondary Outcome: Cerebral Functional Connectivity - Default Mode Network
Description: Functional connectivity is defined as a correlation of the blood oxygenation level dependent (BOLD) signal from each brain network defined by prespecified regions of interest. Whole-brain images were acquired on a GE MR 750 Discovery 3-T scanner using an 8-channel head coil. Functional connectomes were generated using the resting state functional magnetic resonance imaging (fMRI) toolbox. Using the "networks.nii" (with ROIs defined from CONN's ICA analyses of HCP dataset/497 subjects), functional brain networks (e.g., DMN, FPN, SAL, and language) were derived using pairwise BOLD signal correlations, which were then converted to z-scores using Fisher's r-to-z transformation. The DMN, FPN, and SAL were selected as networks of interest due to evidence of the effects of aging and PA on these networks. The language network was selected as a control network.
Time Frame: Baseline and 4 months (follow up)
Population: A subsample of participants in MRI scans. Pre, post change for the Treatment group only was analyzed. Lack of projects funds prohibited analyses of the Control sample (n=4). However, there are plans for this Control sample to be pooled with other Control samples that are part of the same Roybal Center funding to produce a larger sample for analyses.
Measure: Mean (95% Confidence Interval); unit: Average functional connectivity
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 0
Average functional connectivity | -0.0618 [-0.1953 to 0.0716] |

22. Secondary Outcome: Cerebral Functional Connectivity - Frontoparietal Network
Description: as for outcome 21
Time Frame: Baseline and 4 months (follow up)
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: Average functional connectivity
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 0
Average functional connectivity | 0.1013 [0.0037 to 0.1988] |

23. Secondary Outcome: Cerebral Functional Connectivity - Salience Network
Description: as for outcome 21
Time Frame: Baseline and 4 months (follow up)
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: Average functional connectivity
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 0
Average functional connectivity | -0.0422 [-0.1515 to 0.0671] |

24. Secondary Outcome: Cerebral Functional Connectivity - Language Network
Description: as for outcome 21
Time Frame: Baseline and 4 months (follow up)
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: Average functional connectivity
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 10 | 0
Average functional connectivity | 0.0394 [-0.0448 to 0.1237] |

25. Secondary Outcome: Trail Making Test (TMT) Part B
Description: as for outcome 3
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
Seconds | -27.50 [-74.98 to 19.98] | -3.40 [-12.84 to 6.04]

26. Secondary Outcome: Verbal Fluency Test - Fruits and Vegetables
Description: as for outcome 6
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: words
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
words | 0.17 [-2.60 to 2.93] | 2.80 [-2.12 to 7.72]

27. Secondary Outcome: Digit Span Test - Backward
Description: as for outcome 8
Time Frame: Baseline and 4 months (follow up)
Population: Pre to post change within group for participants that completed pre and post data collection.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BAILAMOS© | Control
Number analyzed (Participants) | 12 | 5
score on a scale | 0.33 [-0.45 to 1.11] | -0.20 [-0.75 to 0.36]

ADVERSE EVENTS:
Time Frame: 1 year.
Groups:
- Control While on Waitlist: Randomized to wait list, remained on waitlist for 4 months, received BAILAMOS© program after data collection.
- Control While Participating in BAILAMOS©: Randomized to wait list, received 4-month BAILAMOS© program after data collection.
Arm/Group | BAILAMOS© | Control While on Waitlist | Control While Participating in BAILAMOS©
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 2/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAILAMOS© (N=12) | Control While on Waitlist (N=10) | Control While Participating in BAILAMOS© (N=10)
Headaches (General disorders) | 0 (0) | 2 (2) | 0 (0) — Two participants reported headaches after receiving MRIs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No